CLINICAL TRIAL: NCT04537117
Title: Knowledge, Attitudes and Clinical Practices of Pediatric Dentists Regarding Covid-19
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Maha Moussa Azab, Lecturer of Pediatric Dentistry, Faculty of Dentistry, Fayoum University, Fayoum University
Other Study IDs: pedodontists during Covid-19
Record Dates: First submitted 2020-09-02; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: COVID-19; Pediatric Dentists; Attitudes; Clinical Practices
MeSH Terms: conditions — COVID-19; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric dentists: Pediatric dentists following Facebook groups for pediatric dentists and practicing dentistry nowadays
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — Questionnaire addressing pediatric dentists behaviors and practices during the COVID-19 pandemic

SUMMARY:
This study aims to assess the level of knowledge, attitudes and clinical practices of pediatric dentists regarding COVID-19 pandemic outbreak and evaluate the psychological burden on the dentists and children

DETAILED DESCRIPTION:
Aim: This cross sectional study aims to assess the level of knowledge, attitudes and clinical practices of pediatric dentists regarding COVID-19 pandemic outbreak and evaluate the psychological burden on the dentists and children.

The study population is pediatric dentists recruited through five pediatric dentists Facebook groups. Web-based questionnaire was created using Google forms, structured of multiple-choice questionnaire, and divided into: (demographic, knowledge, practices, and behavior management techniques) sections. Descriptive statistical analysis was used to describe items included in the survey. Numbers and percentages were used to describe categorical data.

ELIGIBILITY:
Inclusion Criteria:

Practicing pediatric dentists working in private practices or institutions

Exclusion Criteria Dentists specialized in other disciplins

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric dentists, practicing during the COVID-19 pandemic
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Responses | 0 days
  Respondents answers to survey questions

CONTACTS AND LOCATIONS:
Overall Officials: Maha M Azab, PhD, Principal Investigator — Fayoum University
Locations (1):
- Fayoum University, Al Fayyum, Egypt